CLINICAL TRIAL: NCT01295359
Title: Impact of a Hospital Physical Therapy Program on Exacerbated Chronic Obstructive Pulmonary Disease Patients: A Randomized Controlled Trial
Brief Title: Impact of a Hospital Physical Therapy Program on Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Valéria Amorim Pires Di Lorenzo, Universidade Federal de São Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPOCexacaminhada
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Walking; Hospital; Exercise Tolerance; Physical Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trained Group (Experimental): This group will receive the usual care of the hospital and a ground walking training program associated with respiratory exercises.
  Interventions: Other: Ground Walking Program
- Usual Care Group (No Intervention): This group will only receive the usual care of the hospital, including physical therapy

INTERVENTIONS:
Other: Ground Walking Program — The patients will walk on a corridor, for 40min, once a day. The speed will be controlled through a metronome, that will be programed to a frequency of steps/min determinated as 80% of the mean frequency of steps performed in six minutes walk test of that day. The 40min will be divided in 3min of walk and 2min of rest, totalizing 24min of exercise and 16min of rest. Furthermore, these patients, in sitting position, will receive orientation to do calm and slow inspirations and expirations, associated with pursed lips expiration. They will try to maintain its Respiratory Rate in 6bpm, during four minutes.
  Other Names: Physical Therapy; Respiratory Rehabilitation
  Arms: Trained Group

SUMMARY:
The Chronic Obstructive Pulmonary Disease is a leading global cause of morbidity and mortality, so it's important to find actions that could improve quality of life and decrease the mortality. The objective of this study is to verify if a ground walking program applied to hospitalized exacerbated COPD patients has effects in quality of life, exercise capacity, airways obstruction, body composition, heart rate variability, quadriceps isometric force and in the "Body-mass index, Airway Obstruction, Dyspnea, Exercise Capacity index" (BODE index). An evaluators-blinded randomized controlled study will be conducted in "Hospital Escola Municipal de São Carlos" where forty patients will be recruited to participate. The volunteers will be randomized in two groups with twenty patients, the usual care group, that will receive only the usual care of the hospital; and the trained group that will receive the same care, but will also participate in a ground walking program associated with respiratory exercises. It will be evaluated, in the start and at the end of the program, the health related and general quality of life and the Barthel index. Daily, the patient will be submitted to the Six Minute Walk Test, to a body composition analysis, to a hand grip test and to a dyspnea assessment, and will be calculated its BODE index. All patients will be invited to a follow up in the 12th and 24th weeks after hospital discharge, when they would receive the same evaluation of the last day in the hospital. All the collected data will be expressed in means and standard deviations or medians and range when appropriated. It will be chosen appropriated tests to compare and correlate them.

ELIGIBILITY:
Inclusion Criteria:

* COPD Patients (FEV1/FVC < 0,70; FEV1 > 30% and < 80%)
* Hospitalized for exacerbation of COPD

Exclusion Criteria:

* Conditions that could restrict walking

  * Skeletal-muscle and joint disturbs
  * Extreme Obesity (BMI > 35kg/m²)
* Heart Failure (New York Heart Association class III and IV)
* Uncontrolled infection (fever > 38ºC and leukocytosis > 10000 cels/dl)
* Need of Invasive Mechanical Ventilation after the beginning of the program
* Previous Diagnosis of:

  * Stroke
  * Epilepsy
* Coagulation disorders (INR > 1,5 or platelets < 50.000/m³)
* Psychiatric Disorders or severe agitation
* Cardiac or respiratory instability
* Oxygen therapy > 3L/min at rest
* Respiratory Rate > 30 breaths/min at rest
* Tachycardia and Bradycardia
* Vasoactive Drugs need

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Change in Exercise Capacity | Daily, as soon as medically appropriated, during the hospitalization
  It will be evaluated through the six minutes walking distance, performed according to ATS rules.
Change in BODE index | Daily, as soon as medically appropriated, during the hospitalization
  The Body-Mass Index, Airways Obstruction, Dyspnea, Exercise Capacity (BODE) index. This is a multidimensional evaluation that includes Forced Expiratory Volume in the first second, Body-Mass Index, 6 Minutes Walking Distance and mMRC score. It is an index to predict mortality.

SECONDARY OUTCOMES:
Change in Perceived Dyspnea | Daily, as soon as medically appropriated, during the hospitalization
  Dyspnea during the six minutes walk test through the BORG CR10 scale
Change in Perceived discomfort in lower limbs | Daily, as soon as medically appropriated, during the hospitalization
  Evaluated during the six minutes walk test through the BORG CR10 scale
Change in Variation in Heart Rate | Daily, as soon as medically appropriated, during the hospitalization
  It will be evaluated the variation in the Heart Rate during the six minutes walk test (Exercise Peak - rest)
Change in the need of oxygen therapy | Daily, as soon as medically appropriated, during the hospitalization
  Will be evaluated the need of oxygen therapy during the six minutes walk test
Change in Handgrip Isometric Force | Daily, as soon as medically appropriated, during the hospitalization
  It will be evaluated through a hand grip dynamometer.
Change in General Quality of Life | first day of the protocol and at the day of discharge
  It will be evaluated through the SF-36 questionnaire
Change in Body Composition | Daily, as soon as medically appropriated, during the hospitalization
  It will be performed through a body composition monitor, evaluating weight, body Fat percentage, Muscle Mass, Basal Metabolic Rate, Bone Mass and Total Body Water Percentage.
Change in Forced Expiratory Volume in the First Second | Daily, as soon as medically appropriated, during the hospitalization
  It will be evaluated through espirometry
Days in hospital | At the discharge
Change in Reported Dyspnea | Daily, as soon as medically appropriated, during the hospitalization
  It will be evaluated through the Modified Medical Research Concil Questionnaire
Change in Heart Rate Variability | first day of the protocol and at the day of discharge
  It will be recorded through a cardiac monitor, and analized in the time and frequency domain, and non-linear analysis.
Quadriceps Isometric Force | first day of the protocol and at the day of discharge
  It will be evaluated through a hand held dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Valéria Amorim Pires Di Lorenzo, PhD, Study Director — Universidade Federal de Sao Carlos; Adriana Sanches Garcia de Araujo, Masters, Principal Investigator — Universidade Federal de Sao Carlos; Juliano Ferreira Arcuri, Especialist, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Hospital Escola Municipal "Dr Horácio Carlos Panepucci, São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Anderson D, Macnee W. Targeted treatment in COPD: a multi-system approach for a multi-system disease. Int J Chron Obstruct Pulmon Dis. 2009;4:321-35. doi: 10.2147/copd.s2999. Epub 2009 Sep 1. PMID 19750192
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Behnke M, Taube C, Kirsten D, Lehnigk B, Jorres RA, Magnussen H. Home-based exercise is capable of preserving hospital-based improvements in severe chronic obstructive pulmonary disease. Respir Med. 2000 Dec;94(12):1184-91. doi: 10.1053/rmed.2000.0949. PMID 11192954
- [Background] Burtin C, Clerckx B, Robbeets C, Ferdinande P, Langer D, Troosters T, Hermans G, Decramer M, Gosselink R. Early exercise in critically ill patients enhances short-term functional recovery. Crit Care Med. 2009 Sep;37(9):2499-505. doi: 10.1097/CCM.0b013e3181a38937. PMID 19623052
- [Background] Burge S, Wedzicha JA. COPD exacerbations: definitions and classifications. Eur Respir J Suppl. 2003 Jun;41:46s-53s. doi: 10.1183/09031936.03.00078002. PMID 12795331
- [Background] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Background] Eaton T, Young P, Fergusson W, Moodie L, Zeng I, O'Kane F, Good N, Rhodes L, Poole P, Kolbe J. Does early pulmonary rehabilitation reduce acute health-care utilization in COPD patients admitted with an exacerbation? A randomized controlled study. Respirology. 2009 Mar;14(2):230-8. doi: 10.1111/j.1440-1843.2008.01418.x. PMID 19272084
- [Background] Faganello MM, Tanni SE, Sanchez FF, Pelegrino NR, Lucheta PA, Godoy I. BODE index and GOLD staging as predictors of 1-year exacerbation risk in chronic obstructive pulmonary disease. Am J Med Sci. 2010 Jan;339(1):10-4. doi: 10.1097/MAJ.0b013e3181bb8111. PMID 19926966
- [Background] Gerardi DA, Lovett L, Benoit-Connors ML, Reardon JZ, ZuWallack RL. Variables related to increased mortality following out-patient pulmonary rehabilitation. Eur Respir J. 1996 Mar;9(3):431-5. doi: 10.1183/09031936.96.09030431. PMID 8730000
- [Background] Kovelis D, Segretti NO, Probst VS, Lareau SC, Brunetto AF, Pitta F. Validation of the Modified Pulmonary Functional Status and Dyspnea Questionnaire and the Medical Research Council scale for use in Brazilian patients with chronic obstructive pulmonary disease. J Bras Pneumol. 2008 Dec;34(12):1008-18. doi: 10.1590/s1806-37132008001200005. English, Portuguese. PMID 19180335
- [Background] Iucif N Jr, Rocha JS. [Study of inequalities in hospital mortality using the Charlson comorbidity index]. Rev Saude Publica. 2004 Dec;38(6):780-6. doi: 10.1590/s0034-89102004000600005. Epub 2004 Dec 10. Portuguese. PMID 15608895
- [Background] MacNee W, Tuder RM. New paradigms in the pathogenesis of chronic obstructive pulmonary disease I. Proc Am Thorac Soc. 2009 Sep 15;6(6):527-31. doi: 10.1513/pats.200905-027DS. PMID 19741262
- [Background] Mathers CD, Boerma T, Ma Fat D. Global and regional causes of death. Br Med Bull. 2009;92:7-32. doi: 10.1093/bmb/ldp028. PMID 19776034
- [Background] Nasis IG, Vogiatzis I, Stratakos G, Athanasopoulos D, Koutsoukou A, Daskalakis A, Spetsioti S, Evangelodimou A, Roussos C, Zakynthinos S. Effects of interval-load versus constant-load training on the BODE index in COPD patients. Respir Med. 2009 Sep;103(9):1392-8. doi: 10.1016/j.rmed.2009.03.003. Epub 2009 Apr 5. PMID 19349153
- [Background] Murphy N, Bell C, Costello RW. Extending a home from hospital care programme for COPD exacerbations to include pulmonary rehabilitation. Respir Med. 2005 Oct;99(10):1297-302. doi: 10.1016/j.rmed.2005.02.033. Epub 2005 Mar 31. PMID 16140230
- [Background] Ong KC, Earnest A, Lu SJ. A multidimensional grading system (BODE index) as predictor of hospitalization for COPD. Chest. 2005 Dec;128(6):3810-6. doi: 10.1378/chest.128.6.3810. PMID 16354849
- [Background] Oxford KL. Elbow positioning for maximum grip performance. J Hand Ther. 2000 Jan-Mar;13(1):33-6. doi: 10.1016/s0894-1130(00)80050-2. PMID 10718220
- [Background] Pinto-Plata VM, Cote C, Cabral H, Taylor J, Celli BR. The 6-min walk distance: change over time and value as a predictor of survival in severe COPD. Eur Respir J. 2004 Jan;23(1):28-33. doi: 10.1183/09031936.03.00034603. PMID 14738227
- [Background] Puhan M, Scharplatz M, Troosters T, Walters EH, Steurer J. Pulmonary rehabilitation following exacerbations of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD005305. doi: 10.1002/14651858.CD005305.pub2. PMID 19160250
- [Background] Seemungal TA, Hurst JR, Wedzicha JA. Exacerbation rate, health status and mortality in COPD--a review of potential interventions. Int J Chron Obstruct Pulmon Dis. 2009;4:203-23. doi: 10.2147/copd.s3385. Epub 2009 Jun 11. PMID 19554195
- [Background] Urbano FL, Pascual RM. Contemporary issues in the care of patients with chronic obstructive pulmonary disease. J Manag Care Pharm. 2005 Jun;11(5 Suppl A):S2-13; quiz S14-6. doi: 10.18553/jmcp.2005.11.s5-a.1. PMID 15934804
- [Background] Vogiatzis I, Nanas S, Roussos C. Interval training as an alternative modality to continuous exercise in patients with COPD. Eur Respir J. 2002 Jul;20(1):12-9. doi: 10.1183/09031936.02.01152001. PMID 12166558
- [Background] Vogiatzis I, Terzis G, Nanas S, Stratakos G, Simoes DC, Georgiadou O, Zakynthinos S, Roussos C. Skeletal muscle adaptations to interval training in patients with advanced COPD. Chest. 2005 Dec;128(6):3838-45. doi: 10.1378/chest.128.6.3838. PMID 16354852